CLINICAL TRIAL: NCT04538690
Title: The Effect of Exercise Therapy on Balance and Pain in Painful Shoulder Disorders
Brief Title: The Effect of Exercise Therapy in Painful Shoulder Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Gizem Ergezen, MSc, Physiotherapist, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-722.02
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Shoulder Pain; Shoulder Disease; Balance; Distorted; Exercise
MeSH Terms: conditions — Shoulder Pain; Motor Activity | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Age and sex matched non interventional, healthy control group
- Exercise Group (Experimental): Individuals who are taken part of shoulder exercises with painful shoulder disorders.
  Interventions: Other: Shoulder Exercises; Other: Electrotherapy

INTERVENTIONS:
Other: Shoulder Exercises — Exercises consist of shoulder range of motion, releasing exercises, strength training, stretching.
  Arms: Exercise Group
Other: Electrotherapy — TENS, US
  Arms: Exercise Group

SUMMARY:
20 adults who applied to the orthopedic clinic with shoulder pain, did not require surgical intervention, were referred to the physiotherapy clinic for treatment; will be evaluated in terms of balance, pain and joint range of motion and then included in the exercise program. 20 adults without pain will be evaluated as the control group and the results will be compared within and between groups. Our hypothesis is that the balance will improve and pain will decrease in individuals after exercise.

DETAILED DESCRIPTION:
20 adults who applied to the orthopedic clinic with shoulder pain, did not require surgical intervention, were referred to the physiotherapy clinic for treatment; will be evaluated in terms of balance, pain and joint range of motion and then included in the exercise program. 20 adults without pain will be evaluated as the control group and the results will be compared within and between groups. Exercises will be applied 3 days a week for 4 weeks, 45-55 minutes by a physiotherapist within the framework of shoulder rehabilitation. In addition, balance exercises will not be given. Balance measurements will be made by the Biodex Balance System, which provides objective data.

ELIGIBILITY:
Inclusion Criteria:

* Having one of the diagnoses of impingement, rotator cuff syndrome, frozen shoulder, biceps tendon,
* Pain severity felt by the patient above-8 according to the Visual Analogue Scale divided into 10 equal intervals,
* Patients who were recommended conservative treatment

Exclusion Criteria:

* Any previous surgical operation,
* Skeletal system fractures or dislocations,
* Other diagnosed orthopedic, neurological or rheumatological diseases, diabetes, neuropathy and pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective Balance Measurement | 4 week
  By Biodex Balance System Stability and Fall Risk, static and dynamic
Pain Intensity | 4 week
  By Visual Analogue Scale scored between 0-10. 0 means no pain and 10 means unbearable pain.

SECONDARY OUTCOMES:
Range of Motion | 4 week
  By Goniometer shoulder range of motion will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)